CLINICAL TRIAL: NCT05264792
Title: Remote Coaching for Supporting the Implementation of Treatment for Depression in Primary Care Facilities in Madhya Pradesh, India: a Cluster Randomized Controlled Trial
Brief Title: Remote Coaching for Supporting the Implementation of Depression Care in Primary Care in Rural India
Acronym: ESSENCE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Sangath (Other); Ministry of Health & Family Welfare, India (Other Government)
Responsible Party: Principal Investigator, John A. Naslund, Instructor of Global Health and Social Medicine, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: U19MH113211-IT; U19MH113211 (NIH)
Record Dates: First submitted 2021-12-30; First posted 2022-03-03 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Depression; Depressive Disorder; Psychological; Noncommunicable Diseases
Keywords: primary care; depression; mental health; implementation; hybrid trial; implementation support strategy
MeSH Terms: conditions — Depression; Depressive Disorder; Noncommunicable Diseases; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study employs a 2-arm parallel cluster-randomized controlled trial design, where the cluster is defined as the Primary Health Centre-Health and Wellness Centre (PHC-HWC). Clusters (14 PHCs-HWCs) are randomly allocated to one of the two implementation support strategies: 1) Routine (existing) implementation support as provided by District Program Management (DPM) team to the facilities (control condition); 2) Enhanced Implementation support consisting of remote coaching provided by the study team in addition to aforementioned Routine Support (intervention condition).
Who Masked: Investigator, Outcomes Assessor
Masking Description: It is not possible to mask collection of implementation outcomes at the facility level or to blind the primary health center staff to arm allocation.
  For patient-level outcomes, outcome assessors and investigators will be masked. Patients who enroll in the study will not be informed about the allocation of their respective facility; therefore, it is unlikely that they would become aware of arm allocation. The study outcome assessors will be blinded to arm allocation of the participants' facilities, and the patient outcome assessments will be conducted at the patient's home or a mutually agreed location, other than the facility. The study team will also ensure separation between the Support Coaching Team delivering the Enhanced Implementation Support strategy and the outcome assessors to avoid any communication that could indicate the arm allocation of participants and facilities.
  The statistician who will analyze the final outcome data will also be blinded to arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine Implementation Support (Active Comparator): All 14 health facilities will continue to receive existing routine implementation support. The facilities allocated to the control arm (n=7) will receive routine implementation support only.
  Interventions: Other: Routine Implementation Support
- Enhanced Implementation Support (Experimental): In addition to routine support, Enhanced Implementation Support will be provided to 7 facilities allocated to the 'intervention arm'.
  Interventions: Other: Enhanced Implementation Support; Other: Routine Implementation Support

INTERVENTIONS:
Other: Enhanced Implementation Support — This support package will include:
  1. one-on-one remote (phone/web-based) technical assistance sessions (every two weeks) between the facility team and the study team Implementation Support Coaches. These sessions will involve a discussion on successes and challenges in integrating depression screening with routine care and developing strategies to improve screening, using the PDSA (Plan Do Study Act) cycle model.
  2. remote peer learning community (peers include ANMs and Nurses who administer screening) through a cross-facility WhatsApp group moderated by the study team Coaching Support Team.
  3. virtual peer learning network conferences (quarterly) moderated by the Coaching Support Team focused on lessons learned in improving depression screening.
  The 9-month intervention duration is informed by the Institute of Healthcare Improvement's Breakthrough Series guidelines.
  Arms: Enhanced Implementation Support
Other: Routine Implementation Support — This support package will include weekly meetings between District and facility teams, to review and discuss mental health performance indicators, such as depression screening rate, refusal rate for PHQ-2 screening, proportion of referrals of screened positive patients from auxiliary nurse midwife (ANM) to Medical Officer, and rates of diagnosis and initiation of treatment of depression. These indicators will be collated and reviewed by the district team as part of existing non-communicable disease (NCD) care indicators. Monthly performance data will be then emailed by the district team to the facilities, in addition to further data submission reminders. Note that these weekly interactions between the district and facility teams does not include the additional PDSA cycle-based coaching support.

SUMMARY:
This cluster-randomized hybrid type-II implementation superiority trial will include 14 rural primary care facilities in Madhya Pradesh, which will implement a collaborative depression care packaged based on the WHO mhGAP program. These 14 facilities will be randomized to receive either 'Enhanced Implementation Support' or the existing 'Routine Implementation Support' control condition to determine if Enhanced Implementation Support is superior to Routine Implementation Support for ensuring successful implementation of the depression care package.

Enhanced Implementation Support consists of remote coaching support and technical assistance. The primary implementation outcome is the proportion of outpatients screened on the PHQ-2 by facility staff. Secondary implementation outcomes will also be collected, including the number of depression cases identified, number of patients with depression referred to the medical officer, number of patients referred to an accepted treatment intervention (i.e., either antidepressant medication or brief psychological intervention), and number of patients who successfully complete treatment at follow up. Secondary patient outcomes will also be collected from patients enrolled in each arm. Patient-level outcomes include the proportion of patients who achieve remission (defined as PHQ-9<5) at 3-month follow up. Additional patient-level outcomes include symptoms of anxiety and functioning.

This trial will develop and test an Enhanced Implementation Support strategy for integrating evidence-based mental health services into primary care facilities. Findings from the trial will inform the need to have external coaching for primary care facilities to meet their depression screening and treatment goals, or if they can achieve these goals via routine system support. This is crucial to inform policymakers, due to severe constraints on mental health budgets for programs in India. Findings can generate insights to inform the scale-up of depression care across other districts in Madhya Pradesh and in India.

DETAILED DESCRIPTION:
Evidence-based clinical interventions exist for depression; however, the gap between those who need treatment and those who receive it (i.e., the care gap) is alarming, with upwards of 90% of individuals not having access to care in India. Integrating evidence-based treatments into primary care is essential for ensuring access to mental health services, and ultimately, bridging the care gap. In India, many of these barriers to implementation have emerged from prior efforts to integrate evidence-based depression care into primary care, such as suboptimal organization and planning, and demands for training of staff on evidence-based interventions.

Implementation research seeks to improve the integration of evidence-based treatments into routine practice through the use of "Implementation Strategies". In a recent review by Wagenaar et al (2020) on implementation strategies for depression care in low- and middle-income countries, it was found that approximately half of these studies were focused on testing revised professional roles, or task-shifting, for depression intervention implementation. In this review, six studies from India examined the integration, acceptability, feasibility and cost of integrating depression care in routine primary care settings, but only one of these studies had a randomized controlled trial design. There is a need to conduct studies with pragmatic designs to examine the effectiveness and cost-effectiveness of integrating evidence-based depression interventions into routine primary care. Moreover, the reviewed studies have scarcely reported on 'adoption' and initial implementation of depression interventions.

This trial aims to address the treatment gap and the structural and contextual factors affecting the optimal implementation of a collaborative care package for depression in primary care settings in Madhya Pradesh, India. Specifically, this study will employ a cluster-randomized controlled design to evaluate whether a 'remote coaching implementation support strategy' compared to 'routine implementation support' can increase rates of screening for depression (i.e., primary implementation outcome). The trial will also assess the successful implementation of the collaborative depression care package via facility-level indicators, including the following secondary implementation outcomes: number of depression cases identified, number of patients with depression referred to the medical officer, number of patients referred to an accepted treatment intervention (i.e., either antidepressant medication or brief psychological intervention), and number of patients who successfully complete treatment at follow up.

Secondary patient outcomes will also be collected from patients enrolled in each arm, including the proportion of patients who achieve remission (defined as PHQ-9<5) at 3-month follow up, given that this reflects a clinically meaningful treatment target. Additional patient-level outcomes include symptoms of anxiety and functioning.

The trial will explore health facility 'readiness' and its relationship with the adoption of the depression care package. Importantly, this trial will employ the routine health facility cadres, such as the auxiliary nurse midwife (ANM) and nurses, primarily for depression screening, and the medical officer (MO) for diagnosis, treatment and referral of cases, and employ routine data collection and management systems. This trial builds on recent health system-level changes in India where screening and management of non-communicable disorders has already been integrated into primary care, creating a template for the integration of evidence-based depression care.

ELIGIBILITY:
Inclusion Criteria:

* Facilities must be primary health centers in Sehore district, Madhya Pradesh, which have been upgraded to "Health and Wellness Center" status offering services for non-communicable disease care, and that have an Accredited Social Health Activist (ASHA) worker linked to the Health and Wellness Center to ensure access to the brief psychological treatment for depression
* Patients must be outpatients seen at these facilities, and must be adults of any gender age ≥18 years
* Patients must screen positive for depression by the ANM/nurse defined as having a PHQ-2 score ≥3.

Exclusion Criteria:

* Facilities that have not been upgraded to Health and Wellness Center and that do not have a linked ASHA worker
* Patients that have significant speech, hearing, language or cognitive impairment impacting their ability to provide informed consent and complete study assessments
* Patients in need of urgent medical or psychiatric attention (e.g., emergency treatment or in-patient admission)
* Patients who do not plan to stay in the study catchment area for at least three months at the time of consent
* Patients who do not understand Hindi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of proportions of persons screened for depression (using PHQ-2) between arms | Baseline to 9-month follow-up
  For the primary implementation outcome, the proportions of outpatients screened on the PHQ-2 by the ANM/nurse will be compared between the study arms. The 2-item Patient Health Questionnaire (PHQ-2) is a widely used brief tool for screening for depression in primary care settings. Scores can range from 0 to 6, with each item scored from 0 (not at all) to 3 (nearly every day). A score of 3 or greater is considered indicative of depressive symptoms. The screenings proportion will be estimated out of the total adult population attending the general outpatient clinics of primary health centers during the trial period. ANMs/nurses will use a Screening Record Register to document the number of patients screened within each facility.

SECONDARY OUTCOMES:
Comparison of number of persons who screen positive for depression on the PHQ-2 (i.e., score ≥3) between arms | Baseline to 9-month follow-up
  Out of the number of patients who are screened for depression using the PHQ-2, the number of outpatients who screen positive for depression (i.e., PHQ-2 score ≥3) will be compared between arms.
Comparison of number of patients with depression (i.e., PHQ-2 score ≥3) who are referred to the Medical Officer (MO) between arms | Baseline to 9-month follow-up
  Out of the number of patients with depression (i.e., PHQ-2 score ≥3), the number who are referred to the Medical Officer (MO) will be compared between arms.
Comparison of number of patients with depression who initiate evidence-based treatment between arms | Baseline to 9-month follow-up
  Out of the number of patients with depression (i.e., PHQ-2 score ≥3) who are referred to the Medical Officer (MO), we will compare the number who initiate treatment, either anti-depressant medication (ADM), brief psychological treatment, or referral to specialty care with a psychiatrist at the District Mental Health Program (DMHP), between arms.
Comparison of number of patients with depression who complete treatment between arms | Baseline to 9-month follow-up
  Out of the number of patients with depression (i.e., PHQ-2 score ≥3) who initiate evidence-based treatment, either anti-depressant medication (ADM), brief psychological treatment, or referral to specialty care with a psychiatrist at the District Mental Health Program (DMHP), the number who complete treatment will be compared between arms. Treatment completion for this trial will be defined as the following: 1) prescribed ADM for 3-month period; 2) attend minimum of 6 sessions of a brief psychological intervention called the Healthy Activity Program (HAP) delivered by ASHAs in the community; and 3) confirmed visit to a specialist mental health provider (i.e., psychiatrist) with the DMHP.
Comparison of proportions of patients who achieve remission (PHQ-9<5) | Baseline and 3-month follow-up
  Out of the patients who screen positive on the PHQ-2 (i.e., score ≥3), the proportion who achieve remission, defined as PHQ-9<5, will be compared between the study arms at 3-month follow up. Patients' PHQ-2 scores collected by the ANM/nurse at the time of screening will be considered as the 'baseline' score for patients who screen positive and consent to participate in the study. The research team will then collect their 3-month follow up PHQ-9 scores (the PHQ-9 is the full 9-item measure of depressive symptoms) at a mutually agreed location. Remission is defined as a PHQ-9 score <5 and is considered a clinically meaningful treatment target in depression care. A 2-week window for collection of follow up assessments from patients will be allowed to accommodate scheduling and other logistics.
Patient Severity of Anxiety assessed with the GAD-7 | Baseline and 3-month follow-up
  Patients' level of anxiety will be measured because it is often co-occurring with depression, yet receives less attention in clinical practice. The outcome assessors will collect the GAD-7, a 7-item self-report scale to screen for symptoms of generalized anxiety disorder. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21, where higher scores indicate more severe anxiety symptoms.
Patient Functional outcomes assessed with the WHODAS 2.0 | Baseline and 3-month follow-up
  The outcome assessors will collect these measures from participants following informed consent at baseline, and then in combination with the primary depression outcome at 3-month follow up at a mutually agreed location. The WHO Disability Assessment Schedule (WHODAS 2.0) consists of 12-items that capture level of functioning across six life domains including cognition, mobility, self-care, getting along, life activities, and participation in society. Each item ranges from 1 (none) to 5 (extreme), with total scores from 12-60. Raw scores are then converted to a summary score ranging from 0 (no disability) to 100 (full disability).

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Tugnawat, Study Director — Sangath; Anant Bhan, MD, Principal Investigator — Sangath
Locations (1):
- Sangath, Bhopal, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) from this trial will be shared with the scientific community according to the National Institute of Mental Health (NIMH) Data Archive Data Sharing terms and conditions. Data will have all direct or indirect identifiable information removed before being submitted to the NIMH Data Archive (NDA). After the trial, the investigators will send de-identified information from participants to NDA. Researchers can access this de-identified data by submitting a request to NIMH. Data sharing with NDA offers no direct benefit to participants, though the information provided to NDA may help researchers around the world treat future mental health challenges so that they have better outcomes. Study participants can choose not to have their de-identified data shared with NDA. These details about data sharing with NDA are described in the participant consent form, and additional information is available at the NDA website.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) will be submitted to the NIMH Data Archive within 12 months after completion of the trial according to the NDA submission schedule and policies.
Access Criteria: There is no plan to restrict access to anonymized data for research purposes. However, access will be provided through the NDA Data Access Committee (DAC). Investigators and institutions seeking data from NDA will be expected to meet data security measures and will be asked to submit a Data Use Certification.
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Bondre AP, Singh A, Tugnawat D, Chandke D, Khan A, Shrivastava R, Lu C, Ramaswamy R, Patel V, Bhan A, Naslund JA. Remote coaching for supporting the implementation of treatment for depression in primary care in Madhya Pradesh, India: protocol for a cluster randomized controlled trial. Front Health Serv. 2024 Sep 24;4:1477444. doi: 10.3389/frhs.2024.1477444. eCollection 2024. PMID 39381591
- [Background] Tugnawat D, Singh A, Anand A, Bondre A, Chandke D, Dhurve P, Joshi U, Khan A, Muke S, Negi B, Nikhare K, Rathore D, Ramaswamy R, Haney JR, Sen Y, Sharma K, Shrivastava R, Verma N, Vishwakarma R, Vishwakarma D, Vorapanya V, Patel V, Bhan A, Naslund JA. ESSENCE: An Implementation Research Program to Scale Up Depression Care in Rural Communities. Psychiatr Serv. 2024 Feb 1;75(2):167-177. doi: 10.1176/appi.ps.202100223. Epub 2023 Oct 31. PMID 37904491